CLINICAL TRIAL: NCT04426032
Title: Predictive Value of Doppler Renal Resistive Index for Prediction of Acute Kidney Injury in Septic Patients in Intensive Care Unit.
Brief Title: Predictive Value of Doppler RSI for Prediction of AKI in Septic Patients in ICU
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mohamed Saleh Ahmed Massoud, Lecturer of Anesthesia and Intensive Care, Ain Shams University
Other Study IDs: FMASU M S 299 / 2020
Record Dates: First submitted 2020-06-09; First posted 2020-06-11 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: Acute Kidney Injury; Sepsis
Keywords: Acute Kidney Injury; Sepsis
MeSH Terms: conditions — Acute Kidney Injury; Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with RRI between 0.6 and 0.7: Normal renal resistive index
  Interventions: Diagnostic Test: Renal Doppler Ultrasound
- Patients with RRI more than 0.7: High renal resistive index
  Interventions: Diagnostic Test: Renal Doppler Ultrasound

INTERVENTIONS:
Diagnostic Test: Renal Doppler Ultrasound — Measurement of Renal resistive index

SUMMARY:
Acute kidney injury (AKI) Diagnosis is based on rising creatinine. Intrarenal vasoconstriction occurs earlier and measuring flow resistance in the renal circulation (Renal Resistive Index (RRI)) could become part of vital organ function assessment using Doppler ultrasound.

The aim of this study is to predict AKI in septic patients in ICU by measuring RRI on admission by comparing two groups of patients, first group with RRI of normal value (0.6-0.7) and the other group with high RRI more than 0.7 and both with normal renal function on admission.

DETAILED DESCRIPTION:
Patients who have criteria of sepsis, with normal renal function on admission will undergo Renal Doppler Ultrasound examination to measure Renal resistive index.

Patients will be divided into 2 groups:

1. Group (A) patients with renal resistive index between 0.6 and 0.7 (normal RRI).
2. Group (B) patients with renal resistive index more than 0.7 (high RRI).

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have criteria of sepsis on admission which include two or more of SIRS which include: (Temperature >38°C or <36°C, Heart rate >90/min, Respiratory rate >20/min or PaCO2 <32mmHg (4.3kPa) and White blood cell count >12000/mm3 or <4000/mm3 or >10% immature bands.) in addition to suspected or confirmed infection.
2. Patients who have normal renal function on admission.

Exclusion Criteria:

1. Currently recovering from an AKI at the time of inclusion and Renal impairment on admission.
2. Patients with obstructive renal failure, renal artery stenosis were excluded from this study.
3. Patients on chemotherapy and/or radiotherapy.
4. Pregnancy.

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: Patients of both sex admitted to ICU, with criteria of sepsis, and normal renal function on admission.
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
incidence of AKI | 1 day at admission
  incidence of AKI related to Renal resistive index.

SECONDARY OUTCOMES:
APACHE III score | 1 day at admission
  Acute Physiology and Chronic Health Evaluation scores. Score range (0 better - 299 worse)
APACHE IV score | 1 day at admission
  Acute Physiology and Chronic Health Evaluation scores. Score range (0 better - 286 worse)
SOFA score | 1 day at admission
  Sequential Organ Failure Assessment (SOFA) score. Score Range (0 better - 24 worse)

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Saleh Ahmed, MD, Study Director — Lecturer of Anesthesia and Intensive Care; Mohammed Saeed Abdelaziz, MD, Study Chair — Professor of Anesthesia and Intensive Care; Mona Refaat Hosney, MD, Study Director — Assistant Professor of Anesthesia and Intensive Care; Ahmed Abdelsattar Abuelmajd, MBBCH, Principal Investigator — Candidate of master degree in general intensive care
Locations (1):
- Ain Shams University Hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
It is not yet known if there will be a plan to make IPD available.